CLINICAL TRIAL: NCT05242653
Title: Comparison of Wound Integrity for Clear Corneal Cataract Incisions: Pressure Versus Stromal Hydration
Brief Title: Comparison of Wound Integrity for Clear Corneal Cataract Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021KYPJ208
Record Dates: First submitted 2022-01-24; First posted 2022-02-16 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cotton swab (Experimental)
  Interventions: Procedure: pressure by a cotton swab
- balanced salt solution (BSS) (Active Comparator)
  Interventions: Procedure: stromal hydration with the balanced salt solution（BSS）

INTERVENTIONS:
Procedure: pressure by a cotton swab — All patients undergo uneventful phacoemulsification by a 2.2 mm temporal transparent corneal incision using Centurion Vision System (Alcon Laboratories, Fort Worth, TX, USA). After the nucleus and cortex are removed, IOL is implanted in the capsular bag. Finally, the clear corneal incision is closed with pressure by a cotton swab.
  Arms: cotton swab
Procedure: stromal hydration with the balanced salt solution（BSS） — All patients undergo uneventful phacoemulsification by a 2.2 mm temporal transparent corneal incision using Centurion Vision System (Alcon Laboratories, Fort Worth, TX, USA). After the nucleus and cortex are removed, IOL is implanted in the capsular bag. Finally, the clear corneal incision is closed with stromal hydration.
  Arms: balanced salt solution (BSS)

SUMMARY:
This is a randomized controlled trial to evaluate the safety and efficacy of two different closing methods for clear corneal cataract incisions

DETAILED DESCRIPTION:
Compared with other incision types , clear corneal incision has the advantages of simple operation, small incision and good healing. It has been widely used in recent decades and has become the most commonly used incision type in phacoemulsification cataract surgery.However, there is no unified standard for the closed method of the clear corneal incision, and some studies have shown that the wound Integrity of clear corneal incision is not well.In the poorly closed incision, the risk of infection increased due to the leakage .Especially in 2.2mm incision, the frequent entry and exit of the instrument reduces the corneal rebound ability at the incision so that the incision is hard to closed. Ensuring wound Integrity for clear corneal cataract incision is the key to the success of cataract surgery.

Clinically closed methods include stromal hydration and suture.The effectiveness of stromal hydration as one of the most commonly used methods has been validated, but also adds additional negative effects. Additionally, the suture extends the operation time and improves the operation cost, and is also accompanied by some complications, which has been less used. Exploring a safe and effective closed method will benefit for most cataract patients.

This study intends to evaluate the safety and efficacy of a closed method that incision is pressed by a cotton swab.The investigators planned to select 130 cataract patients who met the inclusion criteria. The investigators will press the clear corneal incision with a cotton swab in experimental group, while the control group used stromal hydration to close the corneal incision. Wound Integrity, wound leakage, corneal thickness at the incision, keratometric value at the incision, anterior chamber depth and incidence of incision-related descemet membrane detachment were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years old;
2. Nuclear grade is III or IV;
3. Visually significant cataract;
4. The patient is willing and able to complete all necessary follow-ups and examinations.

Exclusion Criteria:

1. Intraoperative or postoperative complications: such as intraoperative posterior capsule rupture, the rupture of zonule, secondary glaucoma, endophthalmitis, etc.;
2. Combined with other eye diseases: such as keratopathy, glaucoma, uveitis, retinopathy, lens dislocation and ocular trauma, etc.;
3. History of intraocular surgery;
4. Severe systemic diseases: such as severe hypertension, diabetes, heart disease, Alzheimer's, Parkinson, etc.;
5. Any condition that the study physician considers to be an impediment to the clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Degree of incision closure | During surgery
  Degree of incision closure is evaluated by intraoperative optical coherence tomography.

SECONDARY OUTCOMES:
Rate of wound leakage | During surgery
  Rate of wound leakage is evaluated by fluorescein sodium.
Corneal thickness | 1 hour after surgery and 1 day after surgery
  Corneal thickness is measured by Casia 2.
Corneal curvature | 1 hour after surgery and 1 day after surgery
  Corneal curvature is measured by Casia 2.
Anterior chamber depth | 1 hour after surgery and 1 day after surgery
  Anterior chamber depth is measured by Casia 2.
Rate of incision-related descemet membrane detachment during surgery | During surgery
  Rate of incision-related descemet membrane detachment is evaluated by intraoperative optical coherence tomography.
Rate of incision-related descemet membrane detachment after surgery | 1 hour after surgery and 1 day after surgery
  Rate of incision-related descemet membrane detachment after surgery is evaluated by Casia 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu Z, Lin H, Jin L, Qu B, Liu J, Zheng Y, He M, Luo L, Liu Y. Swab Pressing vs Stromal Hydration to Prevent Incision Leakage and Transient Collapse of Anterior Chamber in Phacoemulsification: A Randomized Clinical Trial. JAMA Ophthalmol. 2023 Jun 1;141(6):574-581. doi: 10.1001/jamaophthalmol.2023.1491. PMID 37166786